CLINICAL TRIAL: NCT03750721
Title: Staphylococcal Acute Post-Operative Prosthetic Joint Infection Treated With 'DAIR' (Debridement and Implant Retention) And Impact Of Rifampin: A Retrospective Cohort Study In France
Brief Title: Staphylococcal Acute Post-Operative PJI Treated With 'DAIR' And Impact Of Rifampin
Acronym: IPASTAPH
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Principal Investigator, Eugénie MABRUT, Clinical Research Assistant, Hospices Civils de Lyon
Other Study IDs: 18-040
Record Dates: First submitted 2018-08-07; First posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Bone and Joint Infection; Antibiotic Resistant Staphylococcus Aureus Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Role of rifampin in staphylococcal PJI: retrospective cohort study in 4 hospitals : patients with staphylococcal acute post-operative (< 1 month) PJI treated with DAIR in 2011-2016 period
  Interventions: Other: Role of rifampin in staphylococcal PJI

INTERVENTIONS:
Other: Role of rifampin in staphylococcal PJI — the aim is to determine if the dose and the duration of rifampin influenced the prognosis

SUMMARY:
S. aureus and coagulase-negative staphylococci are the most frequent bacteria responsible for PJI (prosthetic joint infection). The aim of this study is to describe the use of rifampicin.

ELIGIBILITY:
Inclusion Criteria:

patients having had acute PJI (i.e. <1 month following the implantation), DAIR with exchange of removal components) due to S. aureus and coagulase-negative staphylococci (2011-2016)

Exclusion Criteria:

None

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: retrospective cohort study in 4 hospitals : patients with staphylococcal acute post-operative (< 1 month) PJI treated with DAIR in 2011-2016 period
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
description of the use of rifampicin : rate of use | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption)
  the aim is to determine how the use of rifampin influence the prognosis in staphylococcal acute post-operative prosthetic joint infection treated with DAIR

SECONDARY OUTCOMES:
rate of failure for treatment using rifampin | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption)
  Treatment failure is defined by local clinical and/or microbiological relapse; and/or need for additional surgery; death of septic origin
rate of adverse event with rifampin | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption)
  Description of adverses events leading to stop the rifampicin

CONTACTS AND LOCATIONS:
Overall Officials: Tristan FERRY, Md,PhD, Principal Investigator — Hospices Civils de Lyon Hôpital de la Croix-Rousse
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided